CLINICAL TRIAL: NCT04706533
Title: Prospective Observational Study Examining Clinical Characteristics, Inflammatory Markers, Treatments and Outcomes of Patients Hospitalized for COVID-19 at the University of Michigan Healthcare System in Ann Arbor
Brief Title: Michigan Medicine COVID-19 Cohort: Clinical Characteristics, Inflammatory Markers and Outcomes of Patients Hospitalized for COVID-19
Acronym: M2C2
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Salim S. Hayek, Assistant Professor of Internal Medicine, University of Michigan
Other Study IDs: HUM00178971
Record Dates: First submitted 2021-01-08; First posted 2021-01-13 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Covid19; Kidney Diseases; Inflammation; SARS-CoV Infection
Keywords: Biomarkers; Outcomes; Inflammation; suPAR; C-reactive protein; Interleukin-6
MeSH Terms: conditions — COVID-19; Kidney Diseases; Inflammation; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum and urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid-19: Patients with confirmed SARS-CoV-2 infection presenting specifically for Covid-19
  Interventions: Diagnostic Test: Biomarkers of inflammation

INTERVENTIONS:
Diagnostic Test: Biomarkers of inflammation — Biomarkers were measured on blood samples collected within 48 hours of admission

SUMMARY:
To better understand the role of inflammation in COVID-19, we established the Michigan Medicine COVID-19 Cohort (M2C2). M2C2 is a funded and ongoing cohort which has currently enrolled over 1500 adult patients (≥18 years) with severe COVID-19 admitted at the University of Michigan. The purpose of M2C2 is to define the in-hospital course of these patients and understand the role of inflammation as a determinant of organ injury and outcomes in COVID-19.

DETAILED DESCRIPTION:
The Michigan Medicine COVID-19 Cohort is a prospective observational cohort study of patients hospitalized specifically for COVID-19 at the University of Michigan Health System in Ann Arbor. Medical records of all consecutive patients with a positive SARS-CoV-2 are reviewed, and patients with confirmed SARS-CoV-2 infection but not primarily admitted for COVID-19 were excluded.

Biologic samples of patients enrolled in M2C2 were collected, and clinical characteristics including in-hospital outcomes were characterized in detail.

Biomarkers measured include, but not be limited to, soluble urokinase plasminogen activator receptor (suPAR), high sensitive C reactive protein (hs-CRP), brain natriuretic protein (BNP), high sensitive troponin T (hsTnT), interleukin 6 (IL-6), osteopontin, a2-antiplasmin.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed SARS-CoV-2 infection
* Hospitalized primarily for the treatment of COVID-19

Exclusion Criteria:

* SARS-CoV-2 positive but hospitalized for non-COVID-19 reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (>18 years) presenting or transferred to the University of Michigan Health System in Ann Arbor
Sampling Method: Non-Probability Sample
Enrollment: 3402 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Death, need for mechanical ventilation or need for dialysis | Total duration of the Covid-19 hospitalization, up to 1 year
  The primary outcome is a composite endpoint, which is defined as the need for mechanical ventilation, the need for dialysis, or in-hospital death.

SECONDARY OUTCOMES:
All-cause death | Total duration of the Covid-19 hospitalization, up to 1 year
Need for mechanical ventilation | Total duration of the Covid-19 hospitalization, up to 1 year
Need for dialysis | Total duration of the Covid-19 hospitalization, up to 1 year

OTHER OUTCOMES:
Length of hospitalization | Total duration of the Covid-19 hospitalization, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Salim Hayek, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data cannot be shared due to consent waiver. Aggregate data and applications for ancillary studies are however available through contacting the Principal Investigator and a application process.

REFERENCES:
- [Background] Azam TU, Shadid HR, Blakely P, O'Hayer P, Berlin H, Pan M, Zhao P, Zhao L, Pennathur S, Pop-Busui R, Altintas I, Tingleff J, Stauning MA, Andersen O, Adami ME, Solomonidi N, Tsilika M, Tober-Lau P, Arnaoutoglou E, Keitel V, Tacke F, Chalkias A, Loosen SH, Giamarellos-Bourboulis EJ, Eugen-Olsen J, Reiser J, Hayek SS; International Study of Inflammation in COVID-19. Soluble Urokinase Receptor (SuPAR) in COVID-19-Related AKI. J Am Soc Nephrol. 2020 Nov;31(11):2725-2735. doi: 10.1681/ASN.2020060829. Epub 2020 Sep 22. PMID 32963090
- [Background] Gupta S, Hayek SS, Wang W, Chan L, Mathews KS, Melamed ML, Brenner SK, Leonberg-Yoo A, Schenck EJ, Radbel J, Reiser J, Bansal A, Srivastava A, Zhou Y, Sutherland A, Green A, Shehata AM, Goyal N, Vijayan A, Velez JCQ, Shaefi S, Parikh CR, Arunthamakun J, Athavale AM, Friedman AN, Short SAP, Kibbelaar ZA, Abu Omar S, Admon AJ, Donnelly JP, Gershengorn HB, Hernan MA, Semler MW, Leaf DE; STOP-COVID Investigators. Factors Associated With Death in Critically Ill Patients With Coronavirus Disease 2019 in the US. JAMA Intern Med. 2020 Nov 1;180(11):1436-1447. doi: 10.1001/jamainternmed.2020.3596. PMID 32667668
- [Background] Gupta S, Coca SG, Chan L, Melamed ML, Brenner SK, Hayek SS, Sutherland A, Puri S, Srivastava A, Leonberg-Yoo A, Shehata AM, Flythe JE, Rashidi A, Schenck EJ, Goyal N, Hedayati SS, Dy R, Bansal A, Athavale A, Nguyen HB, Vijayan A, Charytan DM, Schulze CE, Joo MJ, Friedman AN, Zhang J, Sosa MA, Judd E, Velez JCQ, Mallappallil M, Redfern RE, Bansal AD, Neyra JA, Liu KD, Renaghan AD, Christov M, Molnar MZ, Sharma S, Kamal O, Boateng JO, Short SAP, Admon AJ, Sise ME, Wang W, Parikh CR, Leaf DE; and the STOP-COVID Investigators. AKI Treated with Renal Replacement Therapy in Critically Ill Patients with COVID-19. J Am Soc Nephrol. 2021 Jan;32(1):161-176. doi: 10.1681/ASN.2020060897. Epub 2020 Oct 16. PMID 33067383
- [Background] Hayek SS, Brenner SK, Azam TU, Shadid HR, Anderson E, Berlin H, Pan M, Meloche C, Feroz R, O'Hayer P, Kaakati R, Bitar A, Padalia K, Perry D, Blakely P, Gupta S, Shaefi S, Srivastava A, Charytan DM, Bansal A, Mallappallil M, Melamed ML, Shehata AM, Sunderram J, Mathews KS, Sutherland AK, Nallamothu BK, Leaf DE; STOP-COVID Investigators. In-hospital cardiac arrest in critically ill patients with covid-19: multicenter cohort study. BMJ. 2020 Sep 30;371:m3513. doi: 10.1136/bmj.m3513. PMID 32998872
- [Background] Gupta S, Wang W, Hayek SS, Chan L, Mathews KS, Melamed ML, Brenner SK, Leonberg-Yoo A, Schenck EJ, Radbel J, Reiser J, Bansal A, Srivastava A, Zhou Y, Finkel D, Green A, Mallappallil M, Faugno AJ, Zhang J, Velez JCQ, Shaefi S, Parikh CR, Charytan DM, Athavale AM, Friedman AN, Redfern RE, Short SAP, Correa S, Pokharel KK, Admon AJ, Donnelly JP, Gershengorn HB, Douin DJ, Semler MW, Hernan MA, Leaf DE; STOP-COVID Investigators. Association Between Early Treatment With Tocilizumab and Mortality Among Critically Ill Patients With COVID-19. JAMA Intern Med. 2021 Jan 1;181(1):41-51. doi: 10.1001/jamainternmed.2020.6252. PMID 33080002
- [Background] Flythe JE, Assimon MM, Tugman MJ, Chang EH, Gupta S, Shah J, Sosa MA, Renaghan AD, Melamed ML, Wilson FP, Neyra JA, Rashidi A, Boyle SM, Anand S, Christov M, Thomas LF, Edmonston D, Leaf DE; STOP-COVID Investigators. Characteristics and Outcomes of Individuals With Pre-existing Kidney Disease and COVID-19 Admitted to Intensive Care Units in the United States. Am J Kidney Dis. 2021 Feb;77(2):190-203.e1. doi: 10.1053/j.ajkd.2020.09.003. Epub 2020 Sep 19. PMID 32961244
- [Background] Molnar MZ, Bhalla A, Azhar A, Tsujita M, Talwar M, Balaraman V, Sodhi A, Kadaria D, Eason JD, Hayek SS, Coca SG, Shaefi S, Neyra JA, Gupta S, Leaf DE, Kovesdy CP; STOP-COVID Investigators. Outcomes of critically ill solid organ transplant patients with COVID-19 in the United States. Am J Transplant. 2020 Nov;20(11):3061-3071. doi: 10.1111/ajt.16280. Epub 2020 Sep 15. PMID 32844546
- [Background] Azam TU, Berlin H, Anderson E, Pan M, Shadid HR, Padalia K, O'Hayer P, Meloche C, Feroze R, Michaud E, Launius C, Blakely P, Bitar A, Willer C, Pop-Busui R, Carethers JM, Hayek SS. Differences in Inflammation, Treatment, and Outcomes Between Black and Non-Black Patients Hospitalized for COVID-19: A Prospective Cohort Study. Am J Med. 2022 Mar;135(3):360-368. doi: 10.1016/j.amjmed.2021.10.026. Epub 2021 Nov 16. PMID 34793753
- [Background] Vasbinder A, Anderson E, Shadid H, Berlin H, Pan M, Azam TU, Khaleel I, Padalia K, Meloche C, O'Hayer P, Michaud E, Catalan T, Feroze R, Blakely P, Launius C, Huang Y, Zhao L, Ang L, Mikhael M, Mizokami-Stout K, Pennathur S, Kretzler M, Loosen SH, Chalkias A, Tacke F, Giamarellos-Bourboulis EJ, Reiser J, Eugen-Olsen J, Feldman EL, Pop-Busui R, Hayek SS; ISIC Study Group. Inflammation, Hyperglycemia, and Adverse Outcomes in Individuals With Diabetes Mellitus Hospitalized for COVID-19. Diabetes Care. 2022 Mar 1;45(3):692-700. doi: 10.2337/dc21-2102. PMID 35045184
- [Background] Pan M, Vasbinder A, Anderson E, Catalan T, Shadid HR, Berlin H, Padalia K, O'Hayer P, Meloche C, Azam TU, Khaleel I, Michaud E, Blakely P, Bitar A, Huang Y, Zhao L, Pop-Busui R, Loosen SH, Chalkias A, Tacke F, Giamarellos-Bourboulis EJ, Reiser J, Eugen-Olsen J, Hayek SS; ISIC Group. Angiotensin-Converting Enzyme Inhibitors, Angiotensin II Receptor Blockers, and Outcomes in Patients Hospitalized for COVID-19. J Am Heart Assoc. 2021 Dec 21;10(24):e023535. doi: 10.1161/JAHA.121.023535. Epub 2021 Dec 10. PMID 34889102
- [Background] Wei C, Datta PK, Siegerist F, Li J, Yashwanth S, Koh KH, Kriho NW, Ismail A, Luo S, Fischer T, Amber KT, Cimbaluk D, Landay A, Endlich N, Rappaport J; Michigan Medicine COVID-19 Investigators; Hayek SS, Reiser J. SuPAR mediates viral response proteinuria by rapidly changing podocyte function. Nat Commun. 2023 Jul 21;14(1):4414. doi: 10.1038/s41467-023-40165-5. PMID 37479685
- [Background] Hayek SS, Roderburg C, Blakely P, Launius C, Eugen-Olsen J, Tacke F, Ktena S, Keitel V, Luedde M, Giamarellos-Bourboulis EJ, Luedde T, Loosen SH. Circulating Osteopontin Levels and Outcomes in Patients Hospitalized for COVID-19. J Clin Med. 2021 Aug 30;10(17):3907. doi: 10.3390/jcm10173907. PMID 34501358
- [Background] Vasbinder A, Meloche C, Azam TU, Anderson E, Catalan T, Shadid H, Berlin H, Pan M, O'Hayer P, Padalia K, Blakely P, Khaleel I, Michaud E, Huang Y, Zhao L, Pop-Busui R, Gupta S, Eagle K, Leaf DE, Hayek SS; STOP-COVID Investigatorsdouble dagger. Relationship Between Preexisting Cardiovascular Disease and Death and Cardiovascular Outcomes in Critically Ill Patients With COVID-19. Circ Cardiovasc Qual Outcomes. 2022 Oct;15(10):e008942. doi: 10.1161/CIRCOUTCOMES.122.008942. Epub 2022 Oct 4. PMID 36193749
- [Background] Luo S, Vasbinder A, Du-Fay-de-Lavallaz JM, Gomez JMD, Suboc T, Anderson E, Tekumulla A, Shadid H, Berlin H, Pan M, Azam TU, Khaleel I, Padalia K, Meloche C, O'Hayer P, Catalan T, Blakely P, Launius C, Amadi KM, Pop-Busui R, Loosen SH, Chalkias A, Tacke F, Giamarellos-Bourboulis EJ, Altintas I, Eugen-Olsen J, Williams KA, Volgman AS, Reiser J, Hayek SS; ISIC (International Study of Inflammation in COVID-19) Group. Soluble Urokinase Plasminogen Activator Receptor and Venous Thromboembolism in COVID-19. J Am Heart Assoc. 2022 Sep 20;11(18):e025198. doi: 10.1161/JAHA.122.025198. Epub 2022 Aug 4. PMID 35924778
- [Background] Zhu K, Mukherjee K, Wei C, Hayek SS, Collins A, Gu C, Corapi K, Altintas MM, Wang Y, Waikar SS, Bianco AC, Koch A, Tacke F, Reiser J, Sever S. The D2D3 form of uPAR acts as an immunotoxin and may cause diabetes and kidney disease. Sci Transl Med. 2023 Sep 20;15(714):eabq6492. doi: 10.1126/scitranslmed.abq6492. Epub 2023 Sep 20. PMID 37729431
- [Background] Churpek MM, Gupta S, Spicer AB, Parker WF, Fahrenbach J, Brenner SK, Leaf DE; STOP-COVID Investigators. Hospital-Level Variation in Death for Critically Ill Patients with COVID-19. Am J Respir Crit Care Med. 2021 Aug 15;204(403-411):403-11. doi: 10.1164/rccm.202012-4547OC. PMID 33891529
- [Background] Al-Samkari H, Gupta S, Leaf RK, Wang W, Rosovsky RP, Brenner SK, Hayek SS, Berlin H, Kapoor R, Shaefi S, Melamed ML, Sutherland A, Radbel J, Green A, Garibaldi BT, Srivastava A, Leonberg-Yoo A, Shehata AM, Flythe JE, Rashidi A, Goyal N, Chan L, Mathews KS, Hedayati SS, Dy R, Toth-Manikowski SM, Zhang J, Mallappallil M, Redfern RE, Bansal AD, Short SAP, Vangel MG, Admon AJ, Semler MW, Bauer KA, Hernan MA, Leaf DE; STOP-COVID Investigators. Thrombosis, Bleeding, and the Observational Effect of Early Therapeutic Anticoagulation on Survival in Critically Ill Patients With COVID-19. Ann Intern Med. 2021 May;174(5):622-632. doi: 10.7326/M20-6739. Epub 2021 Jan 26. PMID 33493012
- [Background] Vasquez CR, Gupta S, Miano TA, Roche M, Hsu J, Yang W, Holena DN, Reilly JP, Schrauben SJ, Leaf DE, Shashaty MGS; STOP-COVID Investigators. Identification of Distinct Clinical Subphenotypes in Critically Ill Patients With COVID-19. Chest. 2021 Sep;160(3):929-943. doi: 10.1016/j.chest.2021.04.062. Epub 2021 May 6. PMID 33964301
- [Background] Hsu CM, Gupta S, Tighiouart H, Goyal N, Faugno AJ, Tariq A, Raichoudhury R, Sharma JH, Meyer L, Kshirsagar RK, Jose A, Leaf DE, Weiner DE; STOP-COVID Investigators. Kidney Recovery and Death in Critically Ill Patients With COVID-19-Associated Acute Kidney Injury Treated With Dialysis: The STOP-COVID Cohort Study. Am J Kidney Dis. 2022 Mar;79(3):404-416.e1. doi: 10.1053/j.ajkd.2021.11.004. Epub 2021 Dec 4. PMID 34871701
- See also: Related Info — https://hayek.lab.medicine.umich.edu/research/covid19